CLINICAL TRIAL: NCT04510532
Title: Early Detection of Chemotherapy-related Cardiomyopathy in Patients With Breast Cancer Using Cardiac Magnetic Resonance
Brief Title: Early Detection of CMP in Patients With Breast Cancer Using Cardiac Magnetic Resonance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Ruijin Hospital (Other); Shanghai Fifth People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-08-06R
Record Dates: First submitted 2020-08-07; First posted 2020-08-12 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Chemotherapy Induced Systolic Dysfunction
Keywords: Chemotherapy-induced Cardiomyopathy; pyrotinib/apatinib; Cardiac Magnetic Resonance; Echocardiography
MeSH Terms: conditions — Breast Neoplasms | interventions — Echocardiography; Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Breast Cancer who use pyrotinib: The diagnosis of Breast Cancer was made based on the clinical classification criteria. The subjects were given pyrotinib as having HER2-positive breast cancer with no metastasis.
  Interventions: Diagnostic Test: CMR examination
- Patients with Breast Cancer who use apatinib: The diagnosis of Breast Cancer was made based on the clinical classification criteria. The subjects were given apatinib as having HER2-negative breast cancer with no metastasis.
  Interventions: Diagnostic Test: CMR examination
- Control group: The controls were healthy volunteers who have normal electrocardiographic and echocardiographic results and normal CMR findings
  Interventions: Diagnostic Test: CMR examination

INTERVENTIONS:
Diagnostic Test: CMR examination — After recruiting participants and collecting the baseline information, a CMR scan and a post-processed imaging procedure will be carried on .And the follow-up is planned at 1,6 months after chemotherapy in order to detect the cardiac impairment
  Other Names: Echocardiography; EKG

SUMMARY:
Breast cancer is the most common cancers among women worldwide.Although chemotherapy and surgery have greatly improved the survival rate, most types of chemotherapy have been reported to have varying degrees of cardiotoxicity. The investigators will focus on the cardiotoxicity of pyrotinib and apatinib which belong to the new tyrosine kinase inhibitors in respective chemotherapy among more subjects.

DETAILED DESCRIPTION:
Breast cancer is the most common cancers among women worldwide. Although chemotherapy and surgery have greatly improved the survival rate, most types of chemotherapy have been reported to have varying degrees of cardiotoxicity. We have focused on the field of chemotherapy-related cardiomyopathy. Using the unified magnetic resonance sequences and parameters, effect of chemotherapeutic drugs on the myocardium are studies. Our team's previous pilot study has found that chemotherapy-related cardiomyopathy (CMP) may be predicted within one week after chemotherapy initiation. The specific intervention timing, and the sensitivity and specificity of the early screening indicators are to be explored. At the same time, in patients with human epidermalgrowth factor receptor-2-positive breast cancer, our team observed the change of blood pressure, exercise tolerance and myocardial structure, function and tissue characteristics in patients who used tyrosine kinase inhibitors (pyrotinib and apatinib). This is a supplement to the existing drug knowledge. We are planning to further explore whether it is related to the patient's pre-existing cardiovascular diseases, drug type, dose or dosing. There are no published data addressing the above two research areas. The overall goal is to explore the commonness and specificity of myocardial changes after chemotherapy in breast cancer patients and to predict the development of CMP through multimodality imaging and clinical indices. We aim to propose the CMP time window in respective chemotherapy among more subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years old.
* Invasive breast cancer confirmed by Pathology
* Left ventricular ejection fraction ≥ 50%
* Having not received any prior systemic anti-cancer therapy for advanced disease
* an Eastern Cooperative Oncology Group（ECOG） performance status 0-1
* Providing written informed consent

Inclusion Criteria for Control group:

* Absence of known systemic diseases
* Normal examinations
* Age between 18-70 years old.
* Providing written informed consent

Exclusion Criteria:

* Age <18 years old or >70 years old
* Documented coronary artery disease or prior angiography for coronary artery disease (>50% stenosis).
* Patients with bilateral invasive breast cancers.
* Patients with metastasis of breast cancer confirmed by imaging or pathology
* Patients with standard metallic contraindications to CMR or an estimated glomerular filtration rate < 30 ml/min/1.73 m2.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The subjects were prospectively enrolled into 3 cohorts between October 2019 and July 2020. The cohorts were divided as follows: the breast cancer patients with pyrotinib, the breast cancer patients with apatinib and the control group.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of cardiac condition | change between 1 and 6 months after treatment
  Compose of ejection fraction (%)
Composite endpoint of quantitative fibrosis assessment | change between 1 and 6 months after treatment
  Compose of percentage of extracellular volume (%) and positive rate of late gadolinium enhancement (%).
Exercise tolerance | change between 1 and 6 months after treatment
  6 minutes walking test

CONTACTS AND LOCATIONS:
Overall Officials: Meng Jiang, MD, Study Chair — RenJi Hospital, School of Medicine, Shanghai Jiantong University
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chai Y, Jiang M, Wang Y, Liu Q, Lu Q, Tao Z, Wu Q, Yin W, Lu J, Pu J. Protocol for pyrotinib cardiac safety in patients with HER2-positive early or locally advanced breast cancer-The EARLY-MYO-BC study. Front Cardiovasc Med. 2023 Feb 10;10:1021937. doi: 10.3389/fcvm.2023.1021937. eCollection 2023. PMID 36844736